CLINICAL TRIAL: NCT07004218
Title: Postoperative USG Control and Clinical Follow-up of Massive Rotator Cuff Tendon Ruptures
Status: Enrolling by invitation | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Furkan ARAL, STUDY_CHAİR GAZİ UNİVERSİTY, Gazi University
Other Study IDs: E-77082166-604.01-1134735
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Early Retears and Clinical Outcomes Following Surgical Repair of Massive Rotator Cuff Tears
Keywords: Massive rotator cuff tear; Rotator cuff repair; Retear; Postoperative follow-up; Tendon survivability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to investigate the tendon integrity and clinical outcomes following surgical repair of massive rotator cuff tears. Patients with preoperatively diagnosed massive tears, confirmed by MRI and scheduled for surgery, will be included. Tendon healing will be assessed using ultrasonography at postoperative 2 weeks, 3 months, 6 months, and 12 months. Clinical evaluation will be conducted using standardized scoring systems including ASES, UCLA Shoulder Score, VAS, and thresholds for MCID, SCB, and PASS.

The primary outcome is the rate and timing of retears at 12 months and their correlation with functional recovery. The study also aims to identify prognostic factors affecting tendon survivability, such as age, tear size, and muscle quality. By combining imaging and clinical parameters, this study seeks to contribute to the optimization of postoperative follow-up and rehabilitation strategies in the treatment of massive rotator cuff tears.

DETAILED DESCRIPTION:
This prospective observational study is designed to evaluate tendon healing and functional outcomes following surgical repair of massive rotator cuff tears. The study will be conducted at the Department of Orthopaedics and Traumatology, Gazi University Hospital. Patients aged between 18 and 80 years, diagnosed with massive rotator cuff tears on preoperative MRI and scheduled for surgical intervention, will be included.

Massive tears are defined as full-thickness tears involving two or more rotator cuff tendons and/or showing retraction to the level of the glenoid. Exclusion criteria include irreparable tears, prior shoulder surgery on the affected side, severe glenohumeral arthritis, neurological deficits affecting shoulder function, systemic inflammatory diseases, and inability to comply with follow-up.

Ultrasonographic evaluations of tendon integrity will be performed postoperatively at 2 weeks, 3 months, 6 months, and 12 months. These will be conducted by a radiologist in collaboration with orthopedic residents. Tendon status will be categorized as intact, partial retear, or complete retear. Clinical outcomes will be measured using the American Shoulder and Elbow Surgeons (ASES) Score, the UCLA Shoulder Score, the Visual Analog Scale (VAS), and evaluated in terms of Minimal Clinically Important Difference (MCID), Substantial Clinical Benefit (SCB), and Patient Acceptable Symptom State (PASS).

The primary endpoint is the rate of retear at 12 months and its association with clinical recovery. This study aims to clarify the relationship between early tendon healing and long-term functional outcomes, potentially guiding future management strategies in massive rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a massive rotator cuff tear confirmed by preoperative magnetic resonance imaging (MRI), involving at least two tendons and/or retraction to the glenoid level.

Scheduled for surgical rotator cuff repair at Gazi University Hospital, Department of Orthopaedics and Traumatology.

Ability and willingness to undergo postoperative follow-up and imaging (ultrasound) at 2 weeks, 3 months, 6 months, and 12 months post-surgery.

Ability to provide written informed consent.

No prior surgery on the affected shoulder.

Adequate cognitive and physical capacity to comply with postoperative rehabilitation protocols and outcome assessments.

Exclusion Criteria:

* Previous surgical intervention on the affected shoulder (including rotator cuff repair, shoulder arthroplasty, or arthroscopy).

Irreparable rotator cuff tears determined intraoperatively (e.g., excessive retraction, poor tissue quality).

Presence of advanced glenohumeral osteoarthritis (e.g., Hamada grade ≥ 3).

Neurological disorders affecting shoulder function (e.g., brachial plexopathy, stroke-related hemiparesis).

Systemic inflammatory or rheumatologic diseases (e.g., rheumatoid arthritis, lupus) affecting musculoskeletal function.

Infectious conditions of the shoulder or systemic infection at the time of surgery.

Inability to attend regular follow-ups or comply with the rehabilitation protocol due to psychiatric illness, cognitive impairment, or other medical conditions.

Refusal or inability to provide informed consent.

Poor general health status contraindicating surgery or anesthesia (e.g., ASA IV or higher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients diagnosed with massive rotator cuff tears who are scheduled to undergo surgical repair at the Department of Orthopaedics and Traumatology, Gazi University Hospital. Eligible participants will be between 18 and 80 years of age and will have radiologically confirmed full-thickness rotator cuff tears involving at least two tendons and/or exhibiting tendon retraction to the glenoid level, as identified on preoperative MRI.
  All patients included in the study must be surgical candidates with no prior shoulder operations and must be able to comply with the follow-up schedule and postoperative rehabilitation protocol. The population will be prospectively followed for a minimum of 12 months, with serial clinical and ultrasonographic assessments performed at predefined intervals (2 weeks, 3 months, 6 months, and 12 months postoperatively). Data collected will include demographic characteristics, clinical scores (ASES, UCLA, VAS), and tendon in
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome is tendon integrity at 12 months postoperatively, evaluated by ultrasonography, and its correlation with clinical outcomes including ASES, UCLA, VAS scores, and MCID. Retear presence and timing will also be recorded. | Ultrasonography and clinical evaluations will be conducted at 2 weeks, 3 months, 6 months, and 12 months postoperatively to assess tendon integrity and functional outcomes following rotator cuff repair.
  This prospective observational study aims to evaluate early tendon healing and clinical outcomes following surgical repair of massive rotator cuff tears. Patients diagnosed preoperatively with massive rotator cuff tears via MRI and scheduled for surgery at Gazi University Hospital will be included. Tendon integrity will be assessed through ultrasonography at 2 weeks, 3 months, 6 months, and 12 months postoperatively. Clinical outcomes will be measured using ASES, UCLA Shoulder Score, and VAS, as well as MCID, SCB, and PASS thresholds. The correlation between anatomical healing and functional recovery will be investigated. Patients aged 18-80 years without prior shoulder surgery will be eligible. Exclusion criteria include irreparable tears, neurological disorders, and systemic inflammatory diseases. The primary endpoint is retear rate at 12 months. Data will be collected by orthopedic surgeons and radiologists. This study aims to identify prognostic indicators for tendon survivability

CONTACTS AND LOCATIONS:
Locations (1):
- Gazı University, Çankaya, Ankara, Turkey (Türkiye)